# Effect of Single vs Multiple Prophylactic Antibiotic Doses on Prosthetic Joint Infections Following Primary Total Hip Arthroplasty in Patients with Osteoarthritis at Public and Private Hospitals in Denmark

Statistical Analysis Plan for the Nationwide Cross-Over, Cluster Randomized, Non-inferiority The Pro-Hip-Quality Trial

Authors: Armita A. Abedi<sup>1,2</sup>, Claus Varnum<sup>3,4</sup>, Alma Becic Pedersen<sup>5,6</sup>, Tobias Haugegaard<sup>21</sup>, Kirill Gromov<sup>7</sup>, Jesper Hallas<sup>8</sup>, Pernille Iversen<sup>9</sup>, Thomas Jakobsen<sup>10,11</sup>, Espen Jimenez-Solem<sup>12</sup>, Kristian Kidholm<sup>13</sup>, Anne Kjerulf<sup>14</sup>, Jeppe Lange<sup>15</sup>, Anders Odgaard<sup>16</sup>, Flemming Schønning Rosenvinge<sup>17</sup>, Søren Solgaard<sup>18</sup>, Kim Sperling<sup>19</sup>, Marc Stegger<sup>20</sup>, Robin Christensen<sup>21,22</sup> and Søren Overgaard <sup>1,2</sup>

Trial Registration Number: ClinicalTrials.gov, ID NCT05530551

#### February 6<sup>th</sup>, 2025

#### **Affiliations:**

- 1. Department of Orthopedic Surgery and Traumatology, Copenhagen University Hospital Bispebjerg, Copenhagen, Denmark.
- 2. Department of Clinical Medicine, Faculty of Health and Medical Sciences, University of Copenhagen, Copenhagen, Denmark.
- 3. Department of Orthopedics, Lillebaelt Hospital Vejle, Vejle, Denmark.
- 4. Department of Regional Health Research, University of Southern Denmark, Odense, Denmark.
- 5. Department of Clinical Epidemiology, Aarhus University Hospital, Aarhus, Denmark.
- 6. Department of Clinical Medicine, Aarhus University, Aarhus, Denmark.
- 7. Department of Orthopedic Surgery, Copenhagen University Hospital Hvidovre, Hvidovre, Denmark.
- 8. Department of Public Health, Clinical Pharmacology, Pharmacy, and Environmental Medicine, University of Southern Denmark, Odense, Denmark.
- 9. The Danish Clinical Quality Program-National Clinical Registries (RKKP).
- 10. Department of Orthopedics, Aalborg University Hospital, Denmark.
- 11. Department of Clinical Medicine, Aalborg University Hospital, Denmark.
- 12. Department of Clinical Pharmacology, Copenhagen University Hospital, Bispebjerg and Frederiksberg, Copenhagen, Denmark
- 13. CIMT-Centre for Innovative Medical Technology, Odense University Hospital and University of Southern Denmark, Odense, Denmark.
- 14. Infectious Disease Epidemiology & Prevention, Statens Serum Institut, Copenhagen, Denmark.
- 15. Department of Orthopedic Surgery, Horsens Regional Hospital, Horsens Denmark.
- 16. Department of Orthopaedic Surgery, Centre of Head and Orthopedics and University of Copenhagen. Rigshospitalet Copenhagen, Denmark.
- 17. Department of Clinical Microbiology, Odense University Hospital, 5000 Odense C, Denmark.
- 18. Department of Hip and Knee Surgery, Herlev-Gentofte University Hospital, Hellerup, Denmark.
- 19. Department of Orthopedic Surgery, Næstved Hospital, Næstved, Denmark.
- 20. Department of Bacteria, Parasites and Fungi, Statens Serum Institut, Copenhagen, Denmark.
- 21. Section for Biostatistics and Evidence-Based Research, the Parker Institute, Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark.
- 22. Research Unit of Rheumatology, Department of Clinical Research, University of Southern Denmark, Odense University Hospital, Denmark.

**Principal Investigator: Armita Armina Abedi MD,** Department of Orthopedic Surgery and Traumatology, Copenhagen University Hospital Bispebjerg, Copenhagen, Denmark.

**Study Sponsor:** Søren Overgaard, Professor of Orthopedic Surgery and Traumatology, MD, Dr.med.,
Department of Orthopedic Surgery and Traumatology, Copenhagen University Hospital Bispebjerg, Copenhagen,
Denmark.

Senior Biostatistician and Analysis Support: Robin Christensen (RC), Professor of Biostatistics & Clinical Epidemiology, Section for Biostatistics and Evidence-Based Research, the Parker Institute, Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark and Research Unit of Rheumatology, Department of Clinical Research, University of Southern Denmark, Odense University Hospital, Odense Denmark

**Statistical Analyst: Tobias Haugegaard, MSc; Biostatistics fellow,** Section for Biostatistics and Evidence-Based Research, the Parker Institute, Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark.

**Database Manager: Armita Armina Abedi, MD;** Department of Orthopedic Surgery and Traumatology, Copenhagen University Hospital Bispebjerg, Copenhagen, Denmark.

**Protocol version:** This document has been written based on the information contained in the trial protocol version 1.0, dated 15<sup>th</sup> of June 2022 and the published protocol article from June 21<sup>st,</sup> 2023.

#### **BACKGROUND AND RATIONALE**

A feared complication after total hip arthroplasty (THA) is prosthetic joint infection (PJI), associated with high morbidity and mortality (1-3). Perioperative antimicrobial prophylaxis is a well-established and documented part of standard care to reduce the risk of PJI after THA(4-6). There is however no consensus regarding duration of prophylaxis. Danish national guidelines recommend both one single pre operative dose as well as 24 hours of antibiotic coverage as strategies for antibiotic prophylaxis practice, i.e. a single preoperative dose or a 24 hour coverage using either cloxacillin or the second-generation cephalosporin, cefuroxime(7). The choice of antibiotic agent as well as duration, varies among the different orthopedic departments in Denmark which also reflects the clinical practice internationally.

Antimicrobial resistance poses a persistent and increasing global healthcare problem due to its limited treatment options. In addition, patients may experience systemic toxicity following prolonged use of antibiotics (8-12). Therefore, there is a need for optimizing the use of antibiotics and a reduction would be beneficial, but is should be without risking more infections. No randomized trial has compared one single preoperative dose with 24 hours of antibiotic coverage in THA. This comparison is important to establish best evidence-based practice on antibiotic prophylaxis dosages in the future and combating antimicrobial resistance.

#### **Objectives**

The primary objective of this trial is to compare the effect of single versus multiple prophylactic antibiotic doses administered within 24 hours of primary THA due to osteoarthritis on risk of revision due to PJI within 90 days. The noninferiority of single prophylactic antibiotic would be shown if the upper boundary of the two-sided 95% confidence interval for the Odds Ratio is less than 1.4 for the single prophylactic doses as compared with multiple prophylactic antibiotic doses.

#### **Key secondary objectives**

To compare the effect of single versus multiple prophylactic antibiotic doses administered within 24 hours of primary THA due to osteoarthritis on critical outcomes assessed up to 90 days from surgery: Serious Adverse Events (SAEs), Potential PJI referred to as *PJI-likely*, Length of stay for hospitalization (LOS), Major Adverse Cardiovascular Events, Hospital-treated infections (Other

than those listed above), Community-based antibiotic use, Opioid use, Use of prescribed acetaminophen or non-steroidal anti-inflammatory drugs, Any revision after THA.

#### STUDY METHODS

#### Trial design

The Pro-Hip-Quality OA trial is designed as a pragmatic registry-based, multicenter, open-label, cross-over, cluster-randomized, non-inferiority trial (13-16). The statistical analysis plan (SAP) and trial protocol are reported in accordance with a pragmatic combination of the following CONSORT statements: 'CONSORT for trials conducted using cohorts and routinely collected data (13)', 'Pragmatic Trials (14)' 'Cluster Randomized Trials (15),' 'Randomized Crossover Trials (16)' and 'Noninferiority and Equivalence Randomized trials (17).'This pragmatic registry-based trial design (18) will include cluster randomization of 36 different clinical departments, applying a crossover design. The trial was designed as a nationwide study where all public and private orthopedic departments participated, and all eligible patients were included.

The cluster randomization with embedded cross-over design across 36 clinical centers ensures that each center will administer a specific antibiotic regimen (i.e., either single-dose or multiple-dose) for one year. After the first year, centers will switch to the alternate regimen. This design ensures that each center experiences both interventions over the two-year study, facilitating a balanced comparison between the two treatment protocols. We do not anticipate significant variations in patient characteristics between those enrolled in year 1 and year 2 of the study. This expectation encompasses consistency in key factors: patient demographics (e.g., age, sex), comorbidities, baseline health conditions, disease severity, and treatment indications. Similarly, we do not foresee substantial changes in the clinical setting or study environment over the two years, including protocols for patient recruitment, infection prevention strategies, surgical methods, diagnostic approaches, revisions surgery, or access to healthcare resources. Furthermore, the crossover approach means that the sites are randomized to receive each of the interventions once during separate periods (i.e., study year 1 and 2) acting as their own control group. This may attenuate possible imbalances and variations in site characteristics (19, 20).

Trial registration was performed at ClinicalTrials.gov (NCT05530551) in August 2022. Patient enrolment started at the first departments in September 2022 and the last departments in December 2022. Last patient recruitment was completed on November 30, 2024. The trial has

been approved by The Danish Medicines Agency (Case number: 021091723) and The Committees on Health Research Ethics for The Capital Region of Denmark (VEK) (Case number: 21069108) with the option to opt out of informed consent, based on that both interventions follow standardized clinical practice described in national and international guidelines.

#### Randomization

In this cluster randomized trial, each cluster (any specific department of orthopedic surgery or center; e.g.  $C_1$ ,  $C_2$ ,  $C_3$ , ...,  $C_{36}$ ) is the unit randomized. The outcomes of interest are recorded and analyzed for each participant individually nested within cluster. Participants fulfilling the inclusion criteria will have data treated as planned (organized) conditioning on the local department depending on the year of surgery.

The senior biostatistician was responsible for the randomization process. Each center was allocated based on a code provided by the senior biostatistician responsible and reported to a central database. The randomization and allocation procedure will be known for the given year. To minimize the risk of protocol violations, the steering committee—comprising the study coordinator JSL, the principal investigator AAA, and the sponsor SO, conducted meetings with all departments before the recruitment of the first patient and again after the first year to ensure effective implementation of the cross-over. Local study coordinators have been assigned at each study site prior to study start. The local study investigators consist of a team of an orthopedic surgeon or anesthesiologist and a nurse. The team was responsible for change of the standardized departmental instructions for antibiotic prophylaxis according to randomization, prior to study start. Furthermore, they have been responsible for organization and thorough information of all relevant personnel at the respective study sites. Relevant material has been developed and organized by the authors and distributed to the local study coordinators. Meetings were held in the summer and autumn of 2022. New meetings were done one year later before the cross-over of treatment was planned. Furthermore, any protocol deviations or violations which could occur was reported by the local investigators to the principal investigator and sponsor at 6-month evaluations.

The ITT principle was implemented for all participants allocated to a treatment group  $(X_{\text{Single-dose}})$  and  $X_{\text{Multiple-dose}}$ , respectively). All participants will be followed up, assessed, and analyzed as members of that group. This approach ensures that the results reflect real-world clinical scenarios and maintains the integrity of the randomized design. The study was blinded for the statistical analyst TH but not the patients, investigators, nor departments.

#### Sample size and power calculation

Based on existing Danish national statistics, we anticipated that we will be able to include app. 20,000 eligible individuals having a THA when enrolling consecutively across 36 clinical centers over the two-year period; i.e., that would potentially enable a pragmatic intention-to-treat (ITT) population of up to 10,000 patients in each group (i.e., up to 10,000 individuals exposed to a single-dose antibiotics only).

Choice of the non-inferiority design will enable the deliverance of substantial evidence to change clinical practice if the prevention of PJI with a single dose of prophylactic antibiotic is "no less effective than" antibiotic practices of longer duration (i.e., multiple doses). Members of the Danish orthopedic community have been involved in deciding the potentially increased serious infection rate difference, we are willing to tolerate. Because the sample size is based on the standard flow of THA within the Danish real-world setting, we did not conduct formal power or sample size calculations. Initially, we defined "appreciably worse" serious infection rates and the chances of an erroneously significant result, that is, a false positive, that the medical community will tolerate. The PJI rate in Denmark is between 0.5% and up to 5,1%, (mean 1,2%; 95% CI: 1,0-1,4) varying at departmental level (21). It was decided that we will be willing to tolerate a potentially increased serious infection risk difference of up to 0.1% (1‰ more having a PJI i.e., up to one per thousand).

#### Confidence intervals and p-values

All 95% confidence intervals (95%CIs) and *P*-values will be two sided. We will not apply explicit adjustments for multiplicity, rather we will interpret the key secondary endpoints with caution.

Primary endpoint: If we assume that the PJI risk is similar in the two groups (with 10,000 patients in each) we expect to achieve a precision (narrowness) in the two-sided 95% confidence intervals around the Odds Ratio (OR=1.000) from a Generalized Linear Mixed Model (GLMM), with 95% limits from 0.756 to 1.323; with a Random Effects factor for the 36 individual centers, and Fixed Effect factors for group, period and the interaction between group and period (Group×Period). This was validated through multiple simulations. The same simulations were carried out with a population of 8,000 in each group for sensitivity, resulting in 95 % limits around the Odds Ratio (OR=1.000) from 0.731 to 1.368. Based on the CIs from these simulations, that

have very little variability, and the clinical importance of PJIs, a pragmatic non-inferiority margin should be chosen. Thus, non-inferiority will be shown if the upper limit of the two-sided 95% confidence interval for the odds ratio (derived from the GLMM) is less than 1.4 for the single dose as compared with the multiple doses group.

In addition to the simulations, a bootstrap analysis of 1,000 iterations using the 10,000-patient simulation yielded a 95% confidence interval from 0.763 to 1.374. The proximity of the bootstrap result (1.374) to the proposed margin (1.4) demonstrates that the margin accommodates the variability in the trial design while maintaining sufficient statistical power and clinical importance.

With this approach, we anticipate that the results of this cluster randomized, crossover, non-inferiority trial will generate high-quality evidence that may advance and inform clinical practice on antibiotic prophylaxis dosages in the future.

#### Statistical interim analysis and stopping guidance

No statistical interim analysis was planned on any endpoint (index surgery to 90-day follow-up) between the two groups (i.e., single-dose and multiple-dose) between the two groups (single-dose and multiple-dose), as it was assessed that there would not be sufficient statistical power to conduct a meaningful interim analysis. Performing such an analysis could lead to premature conclusions, posing ethical concerns regarding participant safety and treatment efficacy. Therefore, no interim analysis was planned to uphold our study's scientific integrity and ethical responsibility. The final deadline for patient recruitment was set to 30. November 2024, corresponding to a 2-year study period for the departments that started patient inclusion as of December 1<sup>st</sup>, 2022.

#### Timing of final analysis

The final analysis for the between-group comparison (Single-dose vs. Multiple) for the primary endpoint (index surgery to 90-day follow-up) is planned to be performed after each randomized patient has completed the 90-day follow-up, corresponding to March 1<sup>st</sup>, 2025. The main publication of the trial will be prepared when these data have been received and cleaned. The data is anticipated to be received by May 2025 and the cleaning completed by July 2025. In subsequent manuscripts including exploratory outcomes, secondary longer-term endpoints will be analyzed when the 12 months (corresponding to March 2026) and 60 months (March 2030) has been reached

for all randomized patients followed by preparation of manuscripts with one and five-year outcomes, respectively.

#### Timing of secondary outcome assessments

The time point of the assessment of the primary and secondary outcomes is within 90 days after index surgery: SAES, PJI-likely, LOS, MACE, Hospital-treated infections (other than PJI and PJI-likely), Community-based antibiotic use, use of acetaminophen or non-steroidal anti-inflammatory drugs, and any revision after THA. The outcome of opioid use will be evaluated within 6 months before index surgery and within 90 days after index surgery.

#### STATISTICAL PRINCIPLES

#### Adherence and protocol deviations

This is a pragmatic randomized trial, applying the intention-to-treat (ITT) principle. The main analysis uses the treatment policy estimand, which quantifies the average treatment effect among all the centers who had undergone randomization, regardless of adherence to treatment or crossover (i.e., the intention-to-treat population). The ITT approach ensures that the results reflect real-world clinical practice, accounting for adherence variations and any protocol deviations (22). Deviations from the protocol and adherence will be monitored and documented during data management, but they will not exclude participants from the primary analysis.

#### **Analysis populations**

The primary analyses will be based on the ITT population based on the Full Analysis Set; i.e., all patient's undergoing the prespecified surgery using the antibiotic dose corresponding to the specific cluster and year (cross-over, cluster randomization) (22). Accordingly, participants allocated to a treatment group ( $X_{\text{Single-dose}}$  and  $X_{\text{Multiple-dose}}$ , respectively) will be followed up, assessed, and analyzed as members of that cluster, irrespective of the actual antibiotic regimen used in the specific clinic (i.e., independent of physicians' withdrawals and cross-over phenomena) (23, 24).

#### TRIAL POPULATION

#### Screening data

The total number of patients enrolled during the trial period of 2 years, will be collected and reported according to CONSORT flowchart (see **Figure 1**, Mockup below). Furthermore, the

number of ineligible patients including reason for ineligibility and patients with loss to follow-up will be reported.

#### **Eligibility**

All patients  $\geq$  18 years receiving a primary THA conforming to the following inclusion and exclusion criteria are considered eligible for the trial.

#### Inclusion Criteria:

1. primary and secondary causes of osteoarthritis

#### Exclusion Criteria:

- 1. Patients receiving a primary THA due to either acute or sequelae of proximal femoral or acetabular fractures
- 2. Patients receiving a primary THA due to bone tumor or metastasis

Primary and secondary causes of osteoarthritis include: primary idiopathic arthritis, congenital hip dislocation, Morbus Calvé-Legg-Perthes, epiphysiolysis, dysplasia of the acetabulum, atraumatic caput necrosis, rheumatoid arthritis, Morbus Bechterew, other or other arthritis. Concerning developmental dysplasia, approximately 3% of the patients will have secondary OA due to acetabular dysplasia and 2% due to femoral head necrosis (25).

#### Recruitment

The CONSORT flowchart will comprise number of patients screened, excluded (with reasons) eligible for inclusion in the trial, randomized, receiving their allocated treatment and lost to follow-up (with reasons), included in ITT analysis. The CONSORT flowchart is depicted in Mockup **Figure 1.** 

#### Follow-up

Follow-up are planned based on routine treatment practice and registration in administrative national validated databases and registries. Therefore, participation will not result in additional hospital visits.

Timing of loss to follow-up will be presented in the CONSORT flowchart with numbers and reasons for loss to follow-up given at the 90 days (primary end point) outcome

assessment. Furthermore, the number (with reasons) of loss to follow-up during the course of the trial will be summarized by treatment group.

#### **Baseline patient characteristics**

The following data will be obtained from the patient at baseline: sex, age, height, weight, Bodymass index, American Society of Anesthesiologists classification (ASA), Comorbidity status, socioeconomic status (SES), whether the patient has diabetes (ICD-10 codes E10-E14 from DNPR), year of surgery, antibiotic agent applied as prophylaxis, duration of surgery, type of fixation, type of prosthesis and type of operating room as elaborated in Mockup **Table 1**.

Comorbidity status will be evaluated using the Charlson Comorbidity index Score (CCI) (26). Information about comorbidities will be collected from DNPR (27, 28) after linkage using CRS(29) (27). The CCI score will be calculated based on all primary and secondary diagnoses from hospitalizations and outpatient visits registered as ICD-10 codes in the DNPR over a 10-year period before the primary THA. Although the positive predictive value (PPV) for diagnosis and treatment varies substantially in the DNPR (27), the overall PPV for the 19 Charlson conditions has been found to be 98.0% (30). For each patient that undergoes surgery during the trial period, information on SES will be based on retrieved information on marital status, cohabitation, highest obtained level of education, occupation, family income, and a measure of family liquid assets on the index date retrieved from Statistics Denmark (31). SES will be categorized into the following three domains: educational level, income, and employment status. Educational level will be categorized as low, medium, or high. Low includes no education or high school completed, medium includes vocational education or higher preparatory programs, and high includes a bachelor's or higher degree. Cohabitation status will be classified as living alone, cohabiting, or other. Cohabitation status will be classified as living alone or cohabiting with an adult partner (married, unmarried, or living in multifamily housing). Wealth will be determined using either family income (total in a cohousing family before taxes) or family liquid assets (including cash property value, bank deposits, and securities such as stocks, bonds, and mortgage deeds), depending on the patient's age. For patients aged  $\geq$ 65 years, the standard retirement age in Denmark, family liquid assets will be used, as income may no longer accurately reflect financial status. For patients aged <65 years, family income will be used. Family income at the time of THA is calculated as the average annual pre-tax income in kroner (1 Euro  $\approx 7.5$  Kroner) over the 5 years prior to surgery. Income is classified as above or below the mean for each age group (0-59, 60-69, 70-79, 80+). To account for annual

variations, both measures will be averaged over the 5 years preceding the primary THA. Family income and liquid assets will be each categorized into tertiles (low, medium, and high) for their age and combined into a single wealth variable. Numbers and percentages will be calculated and presented for categorical variables. Means and SD will be computed and presented for continuous variables if data follows a normal distribution. In case continuous variables are not normally distributed, median and interquartile range will be calculated. No tests of statistical significance will be conducted for any baseline characteristic variable. However, imbalances with clinical importance will be noted. The baseline characteristics will be presented as illustrated in Mock-up **Table 1.** 

#### **ANALYSIS**

A flow diagram illustrating dataset construction, including codes where applicable (Appendix A). Every outcome was defined according to specific codes in well-defined registries and databases (Table Appendix B).

#### **Interventions**

Patients will have received either one single dose of preoperative antibiotic (i.e. single dose) or one preoperative antibiotic dose followed by three postoperative dosages administered within the first 24 hours after index surgery (i.e. multiple dose). The dosages and antibiotic agents applied have also been outlined in the protocol article (32) as well as the registration on ClinicalTrials.gov, registration ID NCT05530551 and are the following:

#### **Antibiotic Practice Treatment A and B**

| | | Single-Dose (A) / Multiple-Dose (B) | | Multiple-Dose(B | ) |
|---|---|---|---|---|---|
| Antibiotic | Weight | Preoperative | 6 hours | 12 hours | 18 hours |
| | | dose | postoperative | postoperative | postoperative |
| Cloxacillin i.v. | < 120 kg | 2 g | 1 g | 1 g | 1 g |
| | > 120 kg | 3 g | 2 g | 2 g | 2 g |
| Cefuroxime i.v. | < 120 kg | 1.5 g | 750 mg | 750 mg | 750 mg |
| | > 120 kg | 3 g | 1.5 g | 1.5 g | 1.5 g |

#### Possible transition to oral postoperative antibiotic treatment.

The first postoperative dose of cloxacillin or cefuroxime must be administered intravenously.

| Antibiotic | 12 hours postoperative | 18 hours |
|---|---|---|
| | | postoperative |
| Dicloxacillin oral | 1 g | 1 g |
| Amoxicillin and clavulanic acid oral | 875 mg/125 mg* | 875 mg/125 mg* |

No weight adjustment.

#### Antibiotic Practice in cases of cephalosporin allergy or general beta lactam allergy

| Antibiotic | Weight | Preoperative<br>dose | 8 hours<br>postoperative | 16 hours postoperative |
|---|---|---|---|---|
| Clindamycin i.v. | < 120 kg | 900 mg | 300 mg* | 300 mg* |
| | ≥ 120 kg | 900 mg | 600 mg* | 600 mg* |

<sup>\*</sup>The postoperative dose may be administered orally in the same doses.

#### **Outcome definitions and endpoints**

All Danish residents and citizens are assigned a unique and permanent individual identification number (CPR number) at birth or on immigration. The Civil Registration System number goes through all Danish registries and enables an unambiguous linkage between registries and complete individual level follow-up (27, 28). The primary and key secondary outcomes will be included as endpoints, as illustrated in Mockup Table 2.

*Primary endpoint:* Incidence of PJI: The definition of PJI is based on revision surgery within 90 days of primary THA. Revision surgery is defined as a new surgical intervention the first time after the primary intervention including debridement alone or in combination with complete or partial removal or exchange of any implants.

PJI is defined as the presence of at least one of the following three criteria:

<sup>\*</sup>If the center or region does not have access to amoxicillin and clavulanic acid 875/125 mg, a dose of 1 g / 125 mg (i.e. amoxicillin 500 mg + amoxicillin and clavulanic acid 500 mg/125 mg) may be used.

1. Two or more intraoperative deep-tissue samples of phenotypically indistinguishable bacteria isolated from at least three deep-tissue samples (33)

#### And/or

2. One or more positive intraoperative samples from a closed fluid aspirate AND a biopsy (fluid AND tissue) of phenotypically indistinguishable bacteria isolated (33)

#### And/or

3. A PJI when an indication of deep infection is reported to DHR by the surgeon upon revision surgery (34)

The definition of PJI is based on EBJIS(33), an International Consensus(35), and an algorithm developed to capture cases with PJI using national databases (36). For this trial, the definition of PJI is modified to include the most widely accepted definition of PJI with the main importance set to intraoperative cultures (37, 38). The definition of PJI by EBJIS(33) and the consensus from EBJIS and MSIS classifications of PJI(35) has been modified to exclude histological examination of intraoperative tissue biopsies, erythrocyte sedimentation rate, white blood cell count and biomarker analysis in joint fluid as these analyses are not routinely performed in Denmark. Furthermore, sinus tract communication with the joint or prosthesis visualization will be excluded as these are related to later infections than those occurring within 90 days after index surgery.

The definition has been simplified to allow for the capture of PJI through databases and registries without review of medical files and the modifications are expected only to give minor non-significant changes for the capture of PJI (34, 36). Data will be extracted from DNRP, DHR, MiBA and HAIBA. Positive culture samples (aspirations, tissue biopsies or fluid) must be obtained from the relevant hip joint. As part of standard care, a sample of at least 5 tissue biopsies are obtained at revision surgery. All samples are sent for microbiological analysis at one of ten regional departments of clinical microbiology who have standardized methods for handling of biopsies and culturing. The cumulative proportion of patients remaining PJI-free in the two groups will be presented as illustrated in Mockup Figure 2.

Key secondary endpoints evaluated within 90 days from primary THA

1) Serious Adverse Events (SAEs)

Number of patients with one or more SAEs. SAEs are defined according to the guidelines provided by the International Council for Harmonization of Technical Requirements for Human Use (ICH-GCP) (39). SAE refers to an event involving a significant risk of death or disability of the patient (or their offspring), including, but not limited to, an event that: (1) results in death, (2) is life-threatening – in the investigator's opinion the patient was in immediate risk of death from the adverse event when it appeared, (3) requires hospitalization or prolongs existing hospitalization (4) results in permanent or significant disability. SAEs are recorded from DNPR. The list of ICD10 codes to identify SAEs is listed in Appendix C. This list has been curated to include diagnoses that are considered clinically significant, potentially life-threatening, requiring hospitalization, or resulting in persistent or significant disability/incapacity. To ensure comprehensive coverage and adherence to international standards, any additional codes that meet the criteria for SAEs as defined by the ICH-GCP guidelines will also be included.

#### 2) Potential PJI referred to as PJI-likely

Incidence of potential PJI. PJI-likely is defined as at least one of the two criteria is fulfilled:

A: One single intraoperatively obtained positive culture obtained from reoperation (aspiration fluid OR tissue biopsy) regardless of microorganism

B: One single positive culture obtained from aspiration of synovial fluid regardless of microorganism AND any antibiotic prescriptions (ATC category J01) redeemed

These definitions of PJI-likely are based on a modified version of EBJIS (33) as described previously (see primary outcome) and the study by Milandt *et al.* (40) where first-time revisions with one positive culture were found to have a higher risk of re-revision for PJI.

Cases of PJI-likely, will be captured in HAIBA and MIBA, and registration of antibiotic prescription in NPR. Positive culture samples (aspirations, tissue biopsies or fluid) must be obtained from the relevant hip joint.

#### 3) Length of stay for hospitalization (LOS)

Length of hospital stay (continuous measure [days]) is defined as number of postoperative overnight stays, including transfers to other departments and hospitals within 24 hours. Data on LOS is acquired from DNPR.

#### 4) Major Adverse Cardiovascular Events

Incidence of Major Adverse Cardiovascular Events (MACE). A MACE is defined a priori to include thromboembolic complications including venous thromboembolism, myocardial infarction, atrial fibrillation and stroke based on the diagnostic ICD10 codes listed in Appendix B. VTE is defined a priori as both deep venous thromboembolisms confirmed by compression ultrasound and pulmonary embolism confirmed by spiral computed tomography (CT), ventilation-perfusion scintigraphy or pathological removal of an embolus and based on the following diagnostic ICD10 codes: I26, I80.1-I80.9, I82.1-I82.9, or T81.7B-D. Data will be extracted from DNPR.

#### 5) Hospital-treated infections (Other than those listed above)

Patients with at least one hospital-treated infection are defined as those with first-time hospital admission for a primary or secondary infection diagnosis following discharge from the index THA surgery. Hospital-treated infections are identified from DNPR based on ICD-10 codes listed in Appendix B. The list of infections includes chronic and more rare infections, to detect possible flare-ups in any possible ongoing infections. This outcome does not include infections treated during index admission for arthroplasty surgery.

#### 6) Community-based antibiotic use

Community-based antibiotic use (any community-treated infection or antibiotic use after discharge) is defined as at least one dispensing after discharge from index THA surgery and broad-spectrum antibiotics based on the Anatomical Therapeutic Chemical classification (ATC) codes. All antibiotics in Denmark require prescriptions from a physician. The Danish National Health Service Prescription Database has registered all reimbursed prescriptions from all community pharmacies since 2004. Medications are coded according to the ATC codes listed in Appendix B. All antibiotics in Denmark require prescriptions from a physician and these will be identified using NPR (41). We aim to specifically examine the redemption of ATC code J01E prescriptions within one week following the index operation to capture instances of post-operative urinary tract infections.

#### 7) Opioid use

Patients who received at least one opioid prescription following primary THA surgery. All opioids in Denmark require prescriptions from a physician and these will be identified using NPR (41). The following ATC codes (including all subcodes) are included: N01AH (opioid anesthetics), N02A (opioids), N07BC02 (methadone), and R05DA04 (codeine). Given the lack of a clear definition for opioid users, we defined opioid users as patients who redeemed two opioid prescriptions within six months prior to THA surgery. Conversely, patients who did not redeem two or more opioid prescriptions within this timeframe were classified as opioid naïve. For opioid naïve patients, opioid use post-THA is defined as the redemption of two opioid prescriptions within 90 days following surgery. We assert that two separate redeemed prescriptions confirm actual medication use. We will calculate the treatment dosage based on the number of packages and volume redeemed within 90 days post-surgery. To investigate dosages, all doses will be converted to morphine milligram equivalents using a conversion factor specific to the type of opioid (42, 43).

#### 8) Use of acetaminophen or non-steroidal anti-inflammatory drugs

Patients who received at least one prescription for acetaminophen or nonsteroidal anti-inflammatory drugs (NSAIDs) following THA surgery. Prescriptions of analgesics will be identified using NPR (41). All analgesics in Denmark except 10-tablet packages of acetaminophen / ibuprofen of dose 200mg ibuprofen require prescriptions from a physician. Following ATC codes (including all subcodes) are included M01A (NSAIDs) and N02BE01 (paracetamol). Duration of treatment will be calculated based on the number of packages and volume. Since there is no clear definition of acetaminophen or non-steroidal anti-inflammatory users, we define these users as patients who redeemed two prescriptions within 6 months before THA.

#### 9) Any revision after THA

Revision surgery is defined as a new surgical intervention the first time after the primary intervention, including debridement alone or in combination with complete or partial removal or exchange of any implants. Rate of revision is defined as revision due to any cause within 90 days from primary THA surgery. Any revision will be recorded from DHR and DNPR.

#### **Analysis methods**

All descriptive statistics and statistical analysis will be reported in accordance with the recommendations of the "Enhancing the QUAlity and Transparency Of health Research" (EQUATOR) network (44) and the CONSORT statement (45). Visual inspection (QQ-plot, histograms, and scatterplots) of the standardized residuals from the statistical model will be used to assess the assumption of normality and homogeneity of variances.

The primary analyses will be based on the Intention to Treat (ITT) population, i.e., all patients undergoing the prespecified surgery corresponding to the specific year (cross-over, cluster randomization). Two-sided 95% confidence intervals will be estimated and reported enabling (standard) superiority interpretations. The primary statistical analysis model will be based on a *Generalized Linear Mixed Model*, with a random effects factor applied indexing the clinical center (36 levels: 1, 2, 3, ..., up to 36), a fixed effect will be applied for period (2 levels: 1st and 2nd year, respectively), and antibiotics group (2 levels: Single-dose and Multiple-dose, respectively), as well as the interaction between the two period and antibiotics group (period×group; 4 levels: 2×2 levels). For the primary endpoint: Noninferiority will be shown if the upper limit of the two-sided 95% CI for the odds ratio is less than 1.4 for the single antibiotic doses as compared with multiple doses.

In addition, subgroup analyses will be performed to examine the following known and suspected baseline risk factors for PJI infection will be compared: age ( $\geq$ 65 versus <65 years), sex (male versus female), Anthropometric categories (BMI:  $\geq$ 30 versus <30 kg/m²) as well as morbid obesity (BMI:  $\geq$ 40), and presence of diabetes (with versus without). Additional analyses of the study will assess whether the difference of PJI risk in the two treatment arms differ in specific subsets of patients: femoral stem cementation (antibiotic-loaded bone cement versus bone cement with no antibiotic-load and cementless fixation vs fixation with bone cement) and type of antibiotic (beta-lactam antibiotics versus other). The rationale for these analyses is that we suspect the risk of infection to be different in these subgroups. The pharmacokinetics of the antibiotics might have an impact on the infection rates in the relevant groups. The statistical approach for this evaluation of potential effect modifiers is a test for statistical interaction to evaluate whether the treatment effect varies across levels of the effect modifier (46).

Finally, blinded results from the statistical analyses (single-dose compared to multiple-dose) will be presented to the author group followed by development of two written interpretations. The author group will sign a consensus statement comprising both interpretations prior to the unsealing of the randomization code.(47)

#### Missing data and sensitivity analyses

The main analyses will be based on the data as it appears in the database. Consequently, missing data is handled according to a Missing Completely At Random (MCAR) assumption (48). Conducting sensitivity analyses in a randomized trial assessing the risk of PJIs following a single-dose versus multiple-dose antibiotic prophylaxis is essential to ensure the robustness and credibility of the findings. To evaluate the consistency of the primary endpoint and some or all the key secondary endpoints across various assumptions, missing data will be imputed using best-case, worst-case, best-worst-case, and worst-best-case imputations (49, 50) the results will be combined using Rubin's rule.

#### Additional analyses

Stratified analysis

In secondary analyses, important contextual factors for a binary endpoint will be examined using statistical interaction tests, as proposed by Christensen et al. (46). Known and suspected baseline risk factors for PJI will be evaluated as potential effect modifiers: age group (<65 vs ≥65 years), sex (male vs female), anthropometric category (BMI: <30 vs ≥30 vs > 35 kg/m²) and presence of diabetes (with vs without). Additional analyses of the study will assess whether the difference of PJI risk in the two treatment arms differ in specific subsets of patients: femoral stem cementation (antibiotic-loaded bone cement vs bone cement with no antibiotic-load and cementless fixation vs fixation with bone cement) and type of antibiotic (beta-lactam antibiotics vs other). The rationale for these analyses is that we suspect the risk of infection to be different in these subgroups. The pharmacokinetics of the antibiotics might have an impact on the infection rates in the relevant groups. The statistical approach for this evaluation of potential effect modifiers is a test for statistical interaction to evaluate whether the treatment effect varies across levels of the effect modifier (46). The subgroup analyses will be presented as demonstrated in Mock-up Figure 3A and B. No additional analyses on the primary and key secondary outcomes are planned from baseline to 90-day follow-up.

#### Harms

With regards to safety considerations, this trial will not involve any additional risks of adverse events of the antibiotics exceeding those considered normal for the surgical procedure and administration of antibiotics. Adverse events will be reported following usual practice, from the departments to the Danish Medicines Agency. Antibiotic prophylaxis in this study follows current guidelines for THA surgery. Both cloxacillin, cefuroxime, single dose, and multiple dose regimes are already used as standard practice by Danish surgical centers. The dosage practices are therefore already current standard practices prior to this trial.

As one of the key secondary outcomes, SAEs will be defined in accordance with the "International Conference on Harmonisation-Good Clinical Practice" (ICH-GCP) guidelines.(51) The number (and percentage) of occurrences of all SAEs will be presented for each group. Statistical comparison will be conducted using Risk Differences and Relative Risks as illustrated in Mock-up **Table 3.** 

#### Statistical software

All statistical analyses and calculations will be performed using R version 4.3.2 (2023-10-31 ucrt) with the packages tidyverse, lme4 and emmeans.

#### REFERENCES

- 1. Zmistowski B, Karam JA, Durinka JB, Casper DS, Parvizi J. Periprosthetic joint infection increases the risk of one-year mortality. J Bone Joint Surg Am. 2013;95(24):2177-84.
- 2. Bozic KJ, Ries MD. The impact of infection after total hip arthroplasty on hospital and surgeon resource utilization. J Bone Joint Surg Am. 2005;87(8):1746-51.
- 3. Gundtoft PH, Pedersen AB, Varnum C, Overgaard S. Increased Mortality After Prosthetic Joint Infection in Primary THA. Clin Orthop Relat Res. 2017;475(11):2623-31.
- 4. Doyon F, Evrard J, Mazas F, Hill C. Long-term results of prophylactic cefazolin versus placebo in total hip replacement. Lancet. 1987;1(8537):860.
- 5. van Kasteren ME, Manniën J, Ott A, Kullberg BJ, de Boer AS, Gyssens IC. Antibiotic prophylaxis and the risk of surgical site infections following total hip arthroplasty: timely administration is the most important factor. Clin Infect Dis. 2007;44(7):921-7.
- 6. AlBuhairan B, Hind D, Hutchinson A. Antibiotic prophylaxis for wound infections in total joint arthroplasty: a systematic review. J Bone Joint Surg Br. 2008;90(7):915-9.
- 7. Knæ-alloplastikkirurgi DSfHo. Kort Klinisk Retningslinje, Ortopædisk Kirurgi. Antibiotika profylakse ved alloplastikkirurgi hofte/knæ. 2017:5.
- 8. Branch-Elliman W, O'Brien W, Strymish J, Itani K, Wyatt C, Gupta K. Association of Duration and Type of Surgical Prophylaxis With Antimicrobial-Associated Adverse Events. JAMA Surg. 2019;154(7):590-8.

- 9. Tokarski AT, Karam JA, Zmistowski B, Deirmengian CA, Deirmengian GK. Clostridium difficile is common in patients with postoperative diarrhea after hip and knee arthroplasty. J Arthroplasty. 2014;29(6):1110-3.
- 10. Jacoby GA, Munoz-Price LS. The new beta-lactamases. N Engl J Med. 2005;352(4):380-91.
- 11. Laxminarayan R, Duse A, Wattal C, Zaidi AK, Wertheim HF, Sumpradit N, et al. Antibiotic resistance-the need for global solutions. Lancet Infect Dis. 2013;13(12):1057-98.
- 12. Geneva. WHOGapoar. Global action plan on antimicrobial resistance. Geneva. 2015 09.03.2024. Available from:

https://www.amcra.be/swfiles/files/WHO%20actieplan 90.pdf.

- 13. Kwakkenbos L, Imran M, McCall SJ, McCord KA, Frobert O, Hemkens LG, et al. CONSORT extension for the reporting of randomised controlled trials conducted using cohorts and routinely collected data (CONSORT-ROUTINE): checklist with explanation and elaboration. BMJ. 2021;373:n857.
- 14. Zwarenstein M, Treweek S, Gagnier JJ, Altman DG, Tunis S, Haynes B, et al. Improving the reporting of pragmatic trials: an extension of the CONSORT statement. BMJ. 2008;337:a2390.
- 15. Campbell MK, Piaggio G, Elbourne DR, Altman DG, Group C. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012;345:e5661.
- 16. Dwan K, Li T, Altman DG, Elbourne D. CONSORT 2010 statement: extension to randomised crossover trials. BMJ. 2019;366:l4378.
- 17. Piaggio G, Elbourne DR, Pocock SJ, Evans SJ, Altman DG, Group C. Reporting of noninferiority and equivalence randomized trials: extension of the CONSORT 2010 statement. JAMA. 2012;308(24):2594-604.
- 18. James S, Rao SV, Granger CB. Registry-based randomized clinical trials--a new clinical trial paradigm. Nat Rev Cardiol. 2015;12(5):312-6.
- 19. Arnup SJ, Forbes AB, Kahan BC, Morgan KE, McKenzie JE. Appropriate statistical methods were infrequently used in cluster-randomized crossover trials. (1878-5921 (Electronic)).
- 20. Spence JA-O, Belley-Côté E, Lee SF, Bangdiwala S, Whitlock R, LeManach Y, et al. The role of randomized cluster crossover trials for comparative effectiveness testing in anesthesia: design of the Benzodiazepine-Free Cardiac Anesthesia for Reduction in Postoperative Delirium (B-Free) trial. (1496-8975 (Electronic)).
- 21. Annual reports The Danish Hip Arthorplasy Register 2023. DHR-årsrapport-2019.2024. Available from:
- https://www.sundhed.dk/content/cms/98/4698\_dhr\_aarsrapport\_2023\_udgivet\_2024\_offen tliggjort\_version.pdf.
- 22. Christensen R, Ranstam J, Overgaard S, Wagner P. Guidelines for a structured manuscript: Statistical methods and reporting in biomedical research journals. Acta Orthop. 2023;94:243-9.
- 23. Detry MA, Lewis RJ. The intention-to-treat principle: how to assess the true effect of choosing a medical treatment. Jama. 2014;312(1):85-6.
- 24. Little RJ, D'Agostino R, Cohen ML, Dickersin K, Emerson SS, Farrar JT, et al. The prevention and treatment of missing data in clinical trials. N Engl J Med. 2012;367(14):1355-60.

- 25. Register D. DHR Årsrapport 2021. Annual reports The Danish Hip Arthorplasy Register. 2021. 2021 [Available from: <a href="http://danskhoftealloplastikregister.dk/wp-content/uploads/2022/07/DHR-aarsrapport-2021">http://danskhoftealloplastikregister.dk/wp-content/uploads/2022/07/DHR-aarsrapport-2021</a> Udgivet-2022 offentliggjort-version.pdf.
- 26. Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83.
- 27. Schmidt M, Schmidt SA, Sandegaard JL, Ehrenstein V, Pedersen L, Sørensen HT. The Danish National Patient Registry: a review of content, data quality, and research potential. Clin Epidemiol. 2015;7:449-90.
- 28. Schmidt M, Pedersen L, Sørensen HT. The Danish Civil Registration System as a tool in epidemiology. Eur J Epidemiol. 2014;29(8):541-9.
- 29. Schmidt M, Pedersen L, Sørensen HT. The Danish Civil Registration System as a tool in epidemiology. European Journal of Epidemiology. 2014;29(8):541-9.
- 30. Thygesen SK, Christiansen CF, Christensen S, Lash TL, Sorensen HT. The predictive value of ICD-10 diagnostic coding used to assess Charlson comorbidity index conditions in the population-based Danish National Registry of Patients. BMC Med Res Methodol. 2011;11:83.
- 31. Statistics Denmark [Available from: <a href="https://www.dst.dk/en">https://www.dst.dk/en</a>.
- 32. Abedi AA, Varnum C, Pedersen AB, Gromov K, Hallas J, Iversen P, et al. Effect of single versus multiple prophylactic antibiotic doses on prosthetic joint infections following primary total hip arthroplasty in patients with osteoarthritis at public and private hospitals in Denmark: protocol for a nationwide cross-over, cluster randomised, non-inferiority trial [The Pro-Hip-Quality Trial]. BMJ Open. 2023;13(8):e071487.
- 33. McNally M, Sousa R, Wouthuyzen-Bakker M, Chen AF, Soriano A, Vogely HC, et al. Infographic: The EBJIS definition of periprosthetic joint infection. Bone Joint J. 2021;103-B(1):16-7.
- 34. Gundtoft PH, Pedersen AB, Schonheyder HC, Overgaard S. Validation of the diagnosis 'prosthetic joint infection' in the Danish Hip Arthroplasty Register. Bone Joint J. 2016;98-B(3):320-5.
- 35. Parvizi J, Gehrke T Fau Chen AF, Chen AF. Proceedings of the International Consensus on Periprosthetic Joint Infection. (2049-4408 (Electronic)).
- 36. Gundtoft PH, Overgaard S, Schonheyder HC, Moller JK, Kjaersgaard-Andersen P, Pedersen AB. The "true" incidence of surgically treated deep prosthetic joint infection after 32,896 primary total hip arthroplasties: a prospective cohort study. Acta Orthop. 2015;86(3):326-34.
- 37. Zimmerli W, Trampuz A, Ochsner PE. Prosthetic-joint infections. N Engl J Med. 2004;351(16):1645-54.
- 38. Parvizi J, Gehrke T, Mont MA, Callaghan JJ. Introduction: Proceedings of International Consensus on Orthopedic Infections. The Journal of Arthroplasty. 2019;34(2):S1-S2.
- 39. ICH HARMONISED GUIDELINE. INTEGRATED ADDENDUM TO ICH E6(R1): GUIDELINE FOR GOOD CLINICAL PRACTICE E6(R2) [Internet]. 2016 [cited 12 July 2022]. Available from:
- https://database.ich.org/sites/default/files/E6 R2 Addendum.pdf.
- 40. Milandt NR, Gundtoft PH, Overgaard S. A Single Positive Tissue Culture Increases the Risk of Rerevision of Clinically Aseptic THA: A National Register Study. Clin Orthop Relat Res. 2019;477(6):1372-81.

- 41. Pottegard A, Schmidt SAJ, Wallach-Kildemoes H, Sorensen HT, Hallas J, Schmidt M. Data Resource Profile: The Danish National Prescription Registry. Int J Epidemiol. 2017;46(3):798-f.
- 42. Nielsen S, Degenhardt L, Hoban B, Gisev N. A synthesis of oral morphine equivalents (OME) for opioid utilisation studies. Pharmacoepidemiol Drug Saf. 2016;25(6):733-7.
- 43. Melsen IM, Szépligeti SK, Gundtoft PH, Pedersen AB. Time trends in opioid use for patients undergoing hip fracture surgery in 1997-2018: A Danish population-based cohort study. Eur J Pain. 2024;28(9):1486-96.
- 44. Christensen R, Bliddal H, Henriksen M. Enhancing the reporting and transparency of rheumatology research: a guide to reporting guidelines. Arthritis Res Ther. 2013;15(1):109.
- 45. Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, et al. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55.
- 46. Christensen R, Bours MJL, Nielsen SM. Effect Modifiers and Statistical Tests for Interaction in Randomized Trials. J Clin Epidemiol. 2021;134:174-7.
- 47. Jarvinen TL, Sihvonen R, Bhandari M, Sprague S, Malmivaara A, Paavola M, et al. Blinded interpretation of study results can feasibly and effectively diminish interpretation bias. Journal of clinical epidemiology. 2014;67(7):769-72.
- 48. Christensen R, Ranstam J, Overgaard S, Wagner P. Guidelines for a structured manuscript: Statistical methods and reporting in biomedical research journals. Acta Orthopaedica. 2023;94:243-9.
- 49. Jakobsen JC, Gluud C, Wetterslev J, Winkel P. When and how should multiple imputation be used for handling missing data in randomised clinical trials a practical guide with flowcharts. BMC Med Res Methodol. 2017;17(1):162.
- 50. Liublinska V, Rubin DB. Sensitivity analysis for a partially missing binary outcome in a two-arm randomized clinical trial. Stat Med. 2014;33(24):4170-85.
- 51. International Conference on Harmonisation Expert Working Group. International conference on harmonisation of technical requirements for registration of pharmaceuticals for human use: ICH harmonised tripartite guideline. Guideline for Good Clinical Practice E6 (R1). 1996 [Available from:

https://www.ich.org/fileadmin/Public\_Web\_Site/ICH\_Products/Guidelines/Efficacy/E6/E6\_R1\_Guideline.pdf

Table 1. Baseline Characteristics of the Patients in the ITT population

Single-dose Multiple-dose (N=)(N=)Age — yr Male sex — no. (%) Height — m Weight --- kg Body-mass index — kg/m<sup>2</sup> American Society of Anesthesiologists group, no. (%) 1 2 3 CCI group no. (%) Low Medium 1-2 High 3+ Diabetes no. (%) Antibiotic agent applied no. (%) Cloxacillin Cefuroxime Clindamycin Other Duration of surgery - minutes < 60 61-90 ≥91 Type of fixation no. (%) Antibiotic-loaded bone cement Bone cement with no antibiotic-load Cementless fixation

```
Year of study
```

Year 1, no. (%)

Year 2, no. (%)

Socioeconomic status

Cohabitation

Education

Wealth

Operating room

ĹAF

TAF

<sup>\*</sup> Plus-minus values will be mean  $\pm SD$  unless otherwise indicated.

Table 2. Outcomes in the Intention-to-Treat Population\*

| Outcome | Single-dose | Multiple- | <b>Odds Ratio</b> | †Absolute risk |
|---------|-------------|-----------|-------------------|----------------|
| Outcome | (N = ) | dose | (95% CI) | difference |
| | | (N =) | | (95%CI) |

#### **Primary Outcome**

Prosthetic Joint infection at 90 days, no. (%)

#### **Key Secondary Outcomes**

Serious adverse events (SAE), no. (%)

PJI-likely, no. (%)

Major Adverse Cardiovascular Events, no. (%)

Length of stay (LOS), days

Hospital-treated infections (excluding SSI), no. (%)

Community-based antibiotic use, no. (%)

Opioid use, no. (%)

Use of acetaminophen/non-steroidal anti-inflammatory

drugs, no. (%)

Revision due to any cause, no. (%)

<sup>\*</sup> The primary analyses will be based on the Intention to Treat (ITT) population based on the Full Analysis Set; i.e., all patients undergoing the prespecified surgery using the antibiotic dose corresponding to the specific year (cross-over, cluster randomization). Two-sided 95% confidence intervals will be estimated and reported enabling (standard) superiority interpretations. The primary statistical analysis model will be based on a *Generalized Linear Mixed Model*, with a random effects factor applied indexing the clinical center (36 levels: 1, 2, 3, ..., up to 36), a fixed effect will be applied for period (2 levels: 1st and 2nd year, respectively), and antibiotics group (2 levels: Single-dose and Multiple-dose, respectively), as well as the interaction between the two (period×group; 4 levels: 2×2 levels). Hierarchical models account for variations in baseline risk across clusters (e.g., sites or patient subgroups). †Absolute risk differences and their 95% confidence intervals will be derived from odds ratios and corresponding 95% confidence intervals estimated by the hierarchical model, incorporating the baseline risk in the reference group (multiple-dose). The 95% confidence intervals will not be adjusted for multiplicity and should not be used in place of hypothesis testing.

Table 3. Serious Adverse Events within 90 days within each group. \*

| Events | Single-dose | Multiple-dose | Odds ratio | Absolute risk |
|--------|-------------|---------------|------------|-------------------------|
| | (N = ) | (N =) | (95% CI) | difference <sup>†</sup> |

Serious adverse event — no. (%)

Any infection requiring intravenous antibiotics

Severe allergic reaction

Organ failure

Life-threatening events

Musculoskeletal

Deep infection

Hip dislocation

Femoral fracture

Aseptic loosening

Cardiovascular

Vascular injury

Pulmonary embolism

Deep venous thrombosis

Acute myocardial infarction

Stroke

Nervous system

Nerve injury

Death (All-cause mortality)

Discontinuation due to adverse event(s) — no. (%)

Discontinuation due to serious adverse event(s) — no. (%)

<sup>\*</sup> This table includes all serious adverse events that occurred during the 3month study period, but which did not necessarily have a causal relationship with the treatment administered. An adverse event was classified as serious if it was fatal or life-threatening, required or prolonged inpatient hospitalization, was disabling, resulted in (a congenital anomaly or birth defect), or required medical or surgical intervention to prevent permanent impairment or damage.

<sup>&</sup>lt;sup>†</sup> Absolute risk (single-dose vs. Multiple-dose group) will also be calculated. The 95% confidence intervals will not be adjusted for multiplicity.

FIGURE 1: CONSORT flow-chart.



Figure 2. Kaplan Meier Curve. The cumulative proportion of patients remaining PJI-free in the two groups.



#### Figure 3 Subgroup analyses of the Primary Outcome in the Intention-to-Treat population. The

primary outcome is prosthetic joint infection within 90 days after surgery. The reference group consists of patients assigned to the single-dose group. The confidence intervals for subgroup analyses are not planned to be adjusted for multiplicity and should not be used to infer definitive conclusions about treatment effects. The body-mass index is the weight in kilograms divided by the square of the height in meters. Additional analyses of the risk of PJI 90 days after surgery will assess whether the difference of PJI risk in the two treatment arms differ in specific subsets of patients: femoral stem cementation (antibiotic-loaded bone cement versus bone cement with no antibiotic-load versus cementless fixation) and type of antibiotic (beta-lactam antibiotics versus other). The reference group is patients assigned to single-dose. The rationale for these analyses is that we suspect the risk of infection to be different in these subgroups.



### Appendix A: Flow diagram illustrating dataset construction, including codes where applicable.



Appendix B: Registries, codes, and variables for each outcome

| Outcome | Registry | Codes for Registry |
|---|---|---|
| Primary Outcome: | Danish Hip Arthroplasty | Code for revision for infection in DHR: |
| Prosthetic Joint | Registry (DHR) | |
| infection | | |
| | | DHR: Variable 2: "Revision" |
| | The Hospital Acquired | |
| | Infections Database | HAIBA: Variable "SSI_acute_90 = 0 OR 1", |
| | (HAIBA) | 0 = infection that occurred between 3 and 90 |
| | | days after a planned index operation. |
| | | 1 = infection that occurred between 3 and 90 |
| | The Danish | days after an acute index operation. |
| | Microbiological | MiPA: "Drayedate" corresponding to date or |
| | Database (MiBa) | MiBA: "Prøvedato"=correspondning to date or revision, "Resultat"=positive for microorganism, "Prøvemateriale"=closed fluid aspirate taken |
| | | intraoperatively, "Konklusion på undersøgelse" or<br>"Dyrkningsfund" = phenotypically indistinguishable<br>from bacteria found in tissue biopsy |
| Serious Adverse | The Danish National | Please see Appendix XX for the complete |
| Events | Patient Registry (DNPR) | outline of ICD-10 codes. |
| | The Civil Registration | The civilregistration system: variable: date of |
| | The crimination | death |
| | System | |
| PJI-likely | The Danish | MiBA: "Prøvedato"=between 3 and 90 days after a |
| | Microbiological | planned index operation, "Resultat"=positive for microorganism, "Prøvemateriale"=aspiration of synovial fluid OR closed fluid aspirate taken |

| | Database (MiBa) The Danish National Prescription Registry (NPR) | intraoperatively, "Lokation" = corresponding to THA from index surgery "Undersøgelse" = aspiration with or wihtout imaging guidance or biopsy "Konklusion på undersøgelse" or "Dyrkningsfund" = phenotypically indistinguishable from bacteria found in tissue biopsy From the prescription database (NPR): (ATC |
|---|---|---|
| | | category J01 |
| Length of stay for | The Danish National | From date of index surgery to date of |
| hospitalization | Patient Registry (DNPR) | discharge. |
| Major Adverse | The Danish National | The following ICD.10 codes: |
| Cardiovascular | Patient Registry (DNPR) | |
| Events | | Venous thromboembolism: I26, I80.1 –I80.9, I82 or T81.7 |
| | | Myocardial infarction: I20 – I25 |
| | | Atrial fibrillation: I48.0 -I48.92 |
| | | Stroke: I60.0 - I64.0 |
| Hospital-treated | The Danish National | A20 -A38, A42 -A44, A48 -A49, A65 -A79, |
| infections (Other | Patient Registry (DNPR) | A3, A49.9, A39.4, A40 -A41, B37.7, A32.7, |
| than PJI and PJI- | 5 5 (= 5) | A54.8G, A02.1, A22.7, A26.7, A42.7, A28.2B, |
| likely) | | A06.5, A54.1, B43, D73.3, E06.0A, E23.6A, |
| | | E32.1, G06, G07, H00.0A, H05.0A, H44.0A, |

H60.0, J34.0A, J36, J38.3D, J38.7G, J39.0, J39.1, J39.8A, J85.1, J85.2, J85.3, K04.6, K04.7, K11.3, K12.2, K13.0A, K14.0A, K20.9A, K35.3A, K35.3B, K57.0, K57.2, K57.4, K57.8, K61, K63.0, K65.0, K75.0, K81.0A, K85.8A, L02, L05.0, L05.9, M60.8A, M86.8A, M86.9A, N15.1, N34.0, N41.2, N45.0, N48.2, N49.2A, N61.9A, N61.9B, N70.0A, N70.0B, N71.0A, N73.0A, N73.0B, N73.2A, N73.2B, N73.3A, N73.5A, N73.8A, N73.8C, N75.1, N76.4, N76.8A, Except: A54.1B, B43.0, B43.8, B43.9, K57.0B, K57.0C, K57.2B, K57.2C, K57.4A, K65.0M, K65.0N, K65.0O, K65.0P, A46, H01.0, H03, H60.0, H60.1, H60.2, H60.3, H62, K12.2, K13.0, K61, M72.6, L01, L08, L03, J34.0, L00, L02, L04, L05, L06, L07, L30.3, L73.8, H00, H01.0, H03.0, H03.1, H04.3, H05.0, H06.1, H10, H13.0, H13.1, H15.0, H19.1, H19.2, H22.0, H32.0, H44.0, H44.1, H60, H61.0, H62.0, H62.1, H62.2, H62.3, H65, H66, H67.0, H67.1, H68, H70, H73.0, H75.0, H83.0, H94.0 Except: H60.4, H60.4A, H605, H60.5B, H60.8, H608.A, H65.2, H65.3, H65.4, H65.4C, H66.1, H66.2, H66.3, H68.1, H70.1, H70.8, G00 -07, A80 - A89, G00, G01, G02, G03, A32.1, A39.0, A17.0, A20.3, A87, A54.8D, A02.2C, B37.5, B00.3, B01.0, B02.1, B05.1, B26.1, B38.4, A00 -A09, K35, K37, K57.0, K57.2, K57.4, K57.8, K61, K63.0, K65.0, K65.9, K67, K75.0, K75.1, K80.0, K80.3, K80.4, K81.0, K81.9, K83.0, K85.9, I00 -I02,

| | | , |
|---|---|---|
| | | I30.1, I32.0, I33, I38, I40.0, I39.8, B37.6, J00 - |
| | | J06, J36, J39.0, J39.1, J12 -J18, J20 - J22, |
| | | J44.0, J85.1, J86, J20 -J22, J34.0, J35.0, |
| | | J38.3C, J38.3D, J38.7B, J38.7F, J38.7G, |
| | | <b>Except:</b> J34.0E, J34.0F, J34.0G, J34.0H, N10, |
| | | N11, N12, N15.1, N15.9, N30, N33.0, N34, |
| | | N39.0, N08.0, N13.6, N16.0, N28.8D, N28.8E, |
| | | N28.8F, N29.0, N29.1, Except: N30.1, N30.2, |
| | | N30.4, A50 -A64, N41, N45, N48.1, N48.2, |
| | | N49, N51.1, N51.2, N70 -77, O23, O26.4, |
| | | O41.1, O74.0, O75.3, O85, O86, 088.3, O91, |
| | | O98, M00, M01, M86, M63.0, M63.2, T80.2, |
| | | T81.4, T82.6, T82.7, T83.5, T83.6, T84.5, |
| | | T84.6, T84.7, T85.7, T88.0, T89.9, B90 -B99, |
| | | K04.0, K05.2 |
| | | Codes for specific Hospital-treated infections |
| | | Pneumonia: J12-J18 |
| | | Urinary tract infections N10, N11, N12, N15.1, N15.9, N30, N33.0, N34, N39.0, N08.0, N13.6, N16.0, N28.8D, N28.8E, N28.8F, N29.0, N29.1, Except: N30.1, N30.2, N30.4 |
| Community-based | The Danish National | Narrow spectrum antibiotics: J01CE, J01CF, |
| antibiotic use | Duna animati a u. D. a a i d | J01DB |
| | Prescription Registry | |
| | (NPR) | |
| | | Broad spectrum antibiotics: J01DC, J01DD, |
| | | J01DE, J01DH, J01DI, J01CR, J01CA, J01F. |
| | | J01E, J01MA, J01AA |
| | <u> </u> | |

| Opioid use | The Danish National Prescription Registry (NPR) | Following ATC codes (including all subcodes) are included: N01AH (opioid anesthetics), N02A (opioids), N07BC02 (methadone), and R05DA04 (codeine). |
|---|---|---|
| Use of acetaminophen or non-steroidal anti- inflammatory drugs | The Danish National Prescription Registry (NPR) | Acetaminophen ATC codes: N02BE01 and N02BE51 Non-steroidal anti-inflammatory drug ATC codes: M01A |
| Any revision after THA | Danish Hip Arthroplasty Registry (DHR) and The Danish National Patient Registry (DNPR) | Code for revision for infection in DHR: DHR: Variable 2: "Revision" |

## **Appendix C:** International Classification of Diseases, 10th Revision Diagnosis Codes for Serious Adverse Events

| Serious Adverse Event | ICD-10 Diagnostic Code |
|------------------------------------|------------------------|
| Sepsis | A40 - A41 |
| Shock not elsewhere classifies R67 | R67 |
| Anaphylactic Shock, unspecified | T78.2 |

| Other types of shock included in codes below | <ul> <li>anesthesia (T88.2)</li> <li>anaphylactic (due to): <ul> <li>serum (T80.5)</li> </ul> </li> <li>postoperative (T81.1)</li> <li>traumatic (T79.4)</li> </ul> |
|---|---|
| Staphylococcal scalded skin syndrome | L00 |
| Infectious arthropathies | M00-M03 |
| Osteomyelitis | M86 |
| Injuries to the hip and thigh | S70-S79 |
| Poisoning by drugs, medicaments and | T36 – T50 |
| biological substances | |
| Certain early complications of trauma, not | T79 |
| elsewhere classified | |
| Complications of surgical and medical care, not | T80 – T88 |
| elsewhere classified | |
| Pneumothorax | J93 |
| Respiratory failure, not elsewhere classified | J96 |
| Postprocedural respiratory disorders, not | J95 |
| elsewhere classified | |
| Adult respiratory distress syndrome | J80 |
| Pulmonary oedema | J81 |
| Cardiac arrest | I46 |

| Other forms of heart disease | I30 – I52 |
|---------------------------------------------------------------|-----------|
| Ischemic heart diseases | I20 – I25 |
| Acute and subacute endocarditis | 133 |
| Acute myocarditis | 140 |
| Heart failure | 150 |
| Complications and ill-defined descriptions of heart disease | I51 |
| Pulmonary heart disease and diseases of pulmonary circulation | I26-I28 |
| Arterial embolism and thrombosis | I74 |
| Phlebitis and thrombophlebitis | 180 |
| Portal vein thrombosis | I81 |
| Other venous embolism and thrombosis | 182 |
| Intracranial and intraspinal phlebitis and thrombophlebitis | G08 |
| Postprocedural disorder of circulatory system, unspecified | 197.9 |
| Acute kidney failure | N17 |
| Type 1 diabetes mellitus with diabetic ketoacidosis | E10.1 |

| Type 2 diabetes mellitus with diabetic | E11.1 |
|-------------------------------------------------|-----------|
| ketoacidosis | |
| Other specified diabetes mellitus with diabetic | E13.1 |
| _ | E13.1 |
| ketoacidosis | |
| Stroke | I60-I64 |
| External causes of morbidity and mortality | Y40 – Y84 |
| Acute appendicitis | K35 |
| Acute peritonitis | K65 |
| Perforation of intestine | K63.1 |
| Abscess (perianal, ischiorectal, | K61 |
| intrasphincteric) | |
| Hemoperitoneum | K66.1 |
| Other and unspecified intestinal obstruction | K56.6 |
| Ileus | K56 |
| Hematemesis | K92.0 |
| Melena | 92.1 |
| Gastrointestinal hemorrhage unspecified | 92.2 |
| Acute Pancreatitis | K85 |
| Cholangitis | 83.0 |
| Acute cholecystitis | K81.0 |
| Perforation of gallbladder | K82.2 |
| Abscess of liver | K75.0 |

| Perforation of the esophagus | K22.3 |
|---|---|
| Gastric ulcers with bleeding or perforation | K25.0 to K25.6 |
| Duodenal ulcers with bleeding or perforation | K26.0 to K26.6 |
| Gastrojejunal ulcers with bleeding or | K28.0 to K28.6 |
| perforation | |
| Diverticular disease with perforation, abscess, | K57.0, K57.2, K 57.4, K57.8 |
| or bleeding | |
| Diaphragmatic hernia with obstruction or | K44.0, K44.1 |
| gangrene | |
| Peritonitis | K65 |
| Abscess of intestine | K63.0 |
| Perforation of intestine | K63.1 (non traumatic) |

| Serious Adverse Event | ICD-10 Diagnostic Code |
|-----------------------------|----------------------------------------|
| Surgical site infection | T81.40, T81.41, T81.42, T81.43, T81.49 |
| Venous thromboembolism | I26, I80, T81.7B |
| Cardiac Arrest | I46, I97.12 |
| Acute myocardial Infarction | I21 |
| Stroke | 160 - 164 |
| Pancreatitis | K85 |

| Pneumonia | J13, J14, J15, J16, J17, J18, J85.1, T81-4P |
|---------------------|---------------------------------------------|
| Acute kidney injury | N17 |
| Wound dehiscence | T81.3 |